CLINICAL TRIAL: NCT05941650
Title: To Study the Clinical Effect After Administration of Short-chain Fructooligosaccharides in Women Aged 18 to 65 Years With a Diagnosis of Irritable Bowel Syndrome at the Central State Hospital: A Randomized, Single-blind Study.
Brief Title: To Study the Effect of Short-chain Fructooligosaccharides in Women With Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Chihuahua (Other)
Responsible Party: Principal Investigator, Carolina Martínez Loya, MD, Médico Pasante de Servicio Social, Universidad Autonoma de Chihuahua
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 029C-06/23
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Irritable Bowel Syndrome; Diarrhea- Irritable Bowel Syndrome; Constipation-predominant Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; SC-FOS; Prebiotics
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Prebiotics; Starch

STUDY DESIGN:
Intervention Model Description: Prospective study, randomized single blind clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Chain Fructooligosaccharides Group (Experimental): This group will receive Short-Chain Fructooligosaccharides at a dose of 12 gr. every 24 hours for 10 days, diluted in 250 ml
  Interventions: Dietary Supplement: Short Chain Fructooligosaccharides
- Group (Placebo Comparator): This group will receive Corn Starch as a Placebo control 12 gr. every 24 hours for 10 days, diluted in 250 ml
  Interventions: Other: Corn Starch

INTERVENTIONS:
Dietary Supplement: Short Chain Fructooligosaccharides — The intervention will receive Short-Chain Fructooligosaccharides at a dose of 12 gr. every 24 hours diluted in 250 ml of water.
  Other Names: Prebiotics
  Arms: Short Chain Fructooligosaccharides Group
Other: Corn Starch — This group will receive 12 g of corn starch as a control group.
  Other Names: Placebo
  Arms: Group

SUMMARY:
To evaluate whether there is clinical improvement through the scales (Bristol, IBS severity score, and IBS quality of life) in women with irritable bowel syndrome after administration of SC-FOS (short-chain fructooligosaccharides).

DETAILED DESCRIPTION:
Patients will be selected according to the inclusion and exclusion criteria of the study population for randomization into two groups: one group will be administered short-chain Fructooligosaccharides at a dose of 12 gr. every 24 hours, and the other group will be administered corn starch as a placebo for 10 days.The protocol will be discussed with the patients and/or relatives of the patients, who will understand the consequences and advantages of the study and will sign the informed consent. It should be specified to each patient and/or family member that their participation in the protocol will not generate any extra cost for the administration of SC-FOS, and furthermore, that no reward of any kind will be granted for their participation in the protocol.Once informed consent has been obtained, the preparation (placebo or not) will be delivered to the surgery department of the Central State Hospital. It will come in bags in which the content can be visualized (10 pieces in total, one for each day), numbered according to the folio obtained by the corresponding randomization. It should be emphasized that neither the patient nor the surgery department will know which is a placebo and which contains SC-FOS.There will be a placebo control group and a group that will be administered 12g of SC-FOS, which should be diluted in 250 ml and taken daily for 10 days. Before starting the administration of SC-FOS or placebo, data will be collected on each patient (Bristol Scale, IBS severity score to evaluate severity, IBS quality of life, age, physical activity, drugs, food restriction, time of diagnosis of IBS, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 18 to 65 years
* Irritable Bowel Syndrome diagnosed by Rome Criterion
* Useful enteral feeding

Exclusion Criteria:

* Recent gastrointestinal disease < 2 weeks different to IBS
* Previous consumption of SC-FOS
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Score of IBS-QOL | 10 days
  Score obtained in the questionnaire Irritable Bowel Syndrome - Quality of Life
Score of Bristol Scale | 10 days
  Score obtained by Stool Consistency Bristol Scale
  The seven types of stool are:
  Type 1: Separate hard lumps, like nuts (difficult to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft (average stool) Type 5: Soft blobs with clear cut edges Type 6: Fluffy pieces with ragged edges, a mushy stool (diarrhea) Type 7: Watery, no solid pieces, entirely liquid (diarrhea)
  Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating lack of dietary fiber, and 6 and 7 indicate diarrhoea.
Score of IBS-SSS | 10 days
  Score obtained in the questionnaire Irritable Bowel Syndrome - Severity Scoring System

CONTACTS AND LOCATIONS:
Overall Officials: Luis B Enríquez Sánchez, Study Director — Universidad Autonoma de Chihuahua

IPD SHARING:
Plan to Share IPD: Yes
The data obtained from this research study will be available if requested once the study is finalized.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available for up to five years since completion of the study.
Access Criteria: The request for the data will be by e-mail.